CLINICAL TRIAL: NCT02504658
Title: Mobile Motivation for Health Promotion Among Adolescents
Acronym: BodiMojo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BodiMojo, Inc. (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BodiMojo-R43DK085748; 1R43DK085748-01A1 (NIH)
Record Dates: First submitted 2012-02-02; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes
Keywords: adolescents text messages eating exercise self-efficacy diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Message Group (Experimental): Subjects will set 2 lifestyle goals (exercise and nutrition) and receive health tips and goal status check in messages over 1 month.
  Interventions: Behavioral: Lifestyle text messages
- Control Group (Active Comparator): The control subjects will set 2 lifestyle goals and receive a educational booklet to review.They will take home a copy of the goals they have set. The participants will be also given a 16-page pamphlet from NIDDK "A Guide for Teenagers: Take Charge of Your Health!" to take home to read over. The approximate procedure time will be 20-25 minutes.
  Interventions: Behavioral: Attention Control Group

INTERVENTIONS:
Behavioral: Lifestyle text messages — Throughout the course of the four-week study, the experimental participants will receive one text message each morning related to general nutrition and exercise goals, and an additional "goal status update message" on Monday, Wednesday, and Friday evenings. The goal status update message will ask the participants about the status of attaining their nutrition or physical activity goals. Participants may log their progress toward attaining their goals by using the mobile health dashboard feature on BodiMojo.com from a computer or a web-enabled smartphone to indicate their goal status ("still working on it" or "completed it"). Participants will be encouraged, via the text messages, to look at information on the BodiMojo program found on the Bodimojo.com website.
  Other Names: Experimental
  Arms: Text Message Group
Behavioral: Attention Control Group — Once participants randomized to the control group have completed the baseline assessment, they will be asked to write down two health goals with the RA. The same goals will be suggested for this group as for the Intervention group (see Appendix). They will take home a copy of the goals they have set. The participants will be also given a 16-page pamphlet from NIDDK "A Guide for Teenagers: Take Charge of Your Health!" to take home to read over.
  Other Names: Attention Control
  Arms: Control Group

SUMMARY:
This 4-week pilot study is designed to test the feasibility, adherence, and effectiveness of a cell phone text message program for lifestyle goal setting among adolescents with type 1 or type 2 diabetes. The study entails a small-scale randomized controlled trial with pre-post test of a mobile text message program.

DETAILED DESCRIPTION:
Adolescents with diabetes are a complex target group for health prevention initiatives for a number of developmental reasons, such as drive for autonomy, lack of acknowledgement of long term effects of unhealthy behavior, and high frequency of sedentary behaviors and poor diets (Arnett, 2007). Developing interventions that adolescents find appealing and acceptable is a challenge. An emerging health area referred to as "mobile health" has begun to address these issues by developing innovative uses of basic mobile technologies (Vital Wave/United Nations Foundation, 2009). A recent review of 14 studies, most related to diabetes management (n=10) and preventive behaviors, suggests that mobile phone-delivered interventions have positive short-term behavioral outcomes (Fjedshoe et al., 2009). A number of obesity prevention studies with adults have informed the use of mobile features (e.g., tailored messages or visual display of goal progress) and include mobile applications for adult weight loss (Patrick et al., 2009) and physical activity monitoring for women (Consolvo et al., 2008). Studies targeting children are few. However, one randomized controlled trial of Sweet Talk, a text-messaging system to support young people with diabetes, reported some success (Franklin et al., 2006). In a randomized controlled trial, 126 children with type 1 diabetes were allocated to either conventional insulin therapy, conventional therapy and Sweet Talk (the text message program), or intensive insulin therapy and Sweet Talk. Text messages were tailored to patient's age, sex, and insulin regimen. Compared to conventional treatments, automatic daily text messages (info, tips, support) with weekly reminders about personal goals increased self-efficacy and adherence to diabetes management; overall acceptance rates of Sweet Talk were high (82% felt the program improved self-care; 90% wanted to continue receiving messages). Studies such as these prompted the development of BodiMojo, a mobile phone health application to address healthy nutrition, physical activity, and positive body image. BodiMojo will be tested in the current study with up to 90 adolescents with diabetes to determine feasibility and adherence to lifestyle goals, and to examine changes in self-efficacy. It is hypothesized that the experimental participants will report higher self-efficacy for healthy eating and physical activity, and greater adherence to lifestyle goals, compared to control participants. It is also anticipated that the study procedure, design, and intervention will be found to be feasible. In addition, our group at Joslin has previous experience utilizing text message reminders in adolescents and young adults with type 1 diabetes and demonstrated its acceptability and ease of use (Hanauer, 2006).

Ninety adolescents with diabetes will be recruited to participate in an RCT with a pre- and post-test design to assess feasibility, self-efficacy, and adherence to goal setting. Following informed consent, participants will be randomized to the intervention group or control group and followed for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16-21 years
* Diagnosis of type 1 or type 2 diabetes
* Ownership of a cell phone that supports text messaging
* Intention for continued follow-up care at Joslin
* English-speaking

Exclusion Criteria:

* Current participation in another intervention study or participation in an intervention study in the past 3 months
* Significant developmental or cognitive disorder in the participant that would prevent full participation in the study

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Total Self-Efficacy Score on the Physical Activity and Healthy Food Efficacy Scale for Children | 4 weeks
  The Physical Activity and Healthy Food Efficacy Scale for Children (PAHFE, Perry et al., 2008) is an 18-item instrument designed to assess personal goal-setting self-efficacy and decision-making self-efficacy for physical activity and healthy food choices. This questionnaire was previously used in over 200 adolescents by the co-investigators. An example question is "How sure are you that you can set goals for yourself to eat healthy foods (like fruit & vegetables)?"

SECONDARY OUTCOMES:
Number of text message responses to Goal Setting Question, as a measure of Adherence | 4 weeks
  Adherence will be measured by the frequency of positive or negative responses on status update messages, e.g. "Did you meet your goal today?" [Ans: yes/no]

CONTACTS AND LOCATIONS:
Overall Officials: Tara M Cousineau, PHD, Principal Investigator — BodiMojo, Inc.
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- See also: BodiMojo - Health Promotion portal for teens — http://www.bodimojo.com